CLINICAL TRIAL: NCT07060794
Title: Tafenoquine and DHA-piperaquine (TADORE- Plus)
Acronym: TADORE+
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TADORE+
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tafenoquine plus DHA-Piperaquine (Experimental)
  Interventions: Drug: Tafenoquine
- DHA-Piperaquine (No Intervention)

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine in combination with DHA-piperaquine
  Arms: Tafenoquine plus DHA-Piperaquine

SUMMARY:
A trial designed to determine whether there is a clinically significant drug-drug interaction of tafenoquine with DHA-piperaquine using a control arm with radical cure given at the end of follow up (delayed radical cure).

ELIGIBILITY:
Inclusion Criteria:

* P. vivax peripheral parasitaemia (mono-infection)
* G6PD normal status (G6PD activity ≥70% of the adjusted male median
* as determined by the Standard G6PD (SD Biosensor, ROK))
* Fever (temperature ≥37.5⁰C) or history of fever in the preceding 48 hours
* Age ≥18 years
* Haemoglobin at presentation ≥8g/dl
* Written informed consent.
* Living in the study area and willing to be followed for six months

Exclusion Criteria:

* Danger signs or symptoms of severe malaria
* Pregnant or lactating females
* Regular use of drugs with haemolytic potential
* Known hypersensitivity to any of the study drugs
* History of any psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
incidence risk (time to first event) of any P. vivax parasitaemia | 4 months

IPD SHARING:
Plan to Share IPD: Yes
Submission to WWARN